CLINICAL TRIAL: NCT05557643
Title: PAPR: Psilocybin-assisted Psychotherapy + Mindfulness-Based Stress Reduction (MBSR) for Front-line Healthcare Provider COVID-19 Related Burnout
Brief Title: PAPR: PAP + MBSR for Front-line Healthcare Provider COVID-19 Related Burnout
Acronym: PAPR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Heffter Research Institute (Other); Usona Institute (Other)
Responsible Party: Principal Investigator, Benjamin Lewis, Assistant Professor of Psychiatry, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00152312
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Depression; Burnout, Professional
Keywords: burnout; psilocybin; psychedelic-assisted psychotherapy; healthcare; COVID-19
MeSH Terms: conditions — Depression; Burnout, Professional; Burnout, Psychological; COVID-19 | interventions — Psilocybin; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: 2-arm, randomized, open-label trial for 24 participants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Stress Reduction (MBSR) (Active Comparator): Participants in the MBSR arm will complete an 8-week Mindfulness-Based Stress Reduction Curriculum involving a weekly 2 hour group meeting (either in person or virtual) as well as a 8 hour group mindfulness retreat in week 6-7 of the curriculum.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Mindfulness-Based Stress Reduction (MBSR) + Psilocybin-Assisted Psychotherapy (PAP) (Experimental): Participants in the MBSR + PAP arm will complete an 8-week Mindfulness-Based Stress Reduction Curriculum involving a weekly 2 hour group meeting (either in person or virtual). They will additionally complete a psilocybin-assisted psychotherapy (PAP) intervention that involves three 2-hour group preparatory sessions, a single 8-hour group psilocybin administration session (done in place of the mindfulness retreat), and three 2-hour group integration sessions. All PAP intervention sessions will utilize a 1:1 therapist to participant ratio with an additional lead therapist present.
  Interventions: Drug: Psilocybin; Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is a classic psychedelic of medium duration that is well-tolerated and has a documented safety and efficacy record that makes it uniquely well-suited to the issues that arise in this participant population. Psilocybin has been described as an 'existential medicine' given patient testimonials as to its acute and lasting effects on interpersonal connection, ability to more deeply engage with meaningful activities and relationships, dramatic reductions in fear of death, and a renewed sense of well-being.
  Arms: Mindfulness-Based Stress Reduction (MBSR) + Psilocybin-Assisted Psychotherapy (PAP)
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Mindfulness-Based Stress Reduction (MBSR) is a well-established evidence-based mindfulness training program initially developed by Jon Kabat-Zinn that has been shown to reduce symptoms of depression, anxiety, and burnout. The 8-week MBSR curriculum provides training in formal meditation practices including body scan techniques, mindfulness meditation, and yoga. Mindfulness can be understood as the non-judgmental acceptance and investigation of present experience, including body sensations, internal mental states, thoughts, emotions, impulses and memories, in order to reduce suffering or distress and to increase well-being.

SUMMARY:
This project is an open-label randomized study looking at an 8-week Mindfulness-Based Stress Reduction (MBSR) curriculum vs. an 8-week MBSR curriculum + a group psilocybin-assisted psychotherapy intervention for frontline healthcare providers struggling with symptoms of depression and burnout associated with the SARS-CoV-2 pandemic.

Following consenting and enrollment a total of 24 participants will be randomized to receive either an 8-week MBSR curriculum or the same 8-week MBSR curriculum + a group psilocybin-assisted psychotherapy intervention. The group psilocybin-assisted psychotherapy intervention will involve 3 group preparatory sessions (2 hours each), a single 8 hour group psilocybin administration session with a 1:1 therapist to participant ratio (25mg psilocybin dose), and 3 group integration sessions (2 hours each).

ELIGIBILITY:
Inclusion Criteria:

___ Participants must be physicians or nurses with at least 1 month of frontline clinical experience during the COVID pandemic.

Yes/No Eligibility Questions (Response of "no" = subject ineligible)

* PHQ-9 score ≥ 10 and meet criteria for a DSM-5 depressive disorder (including adjustment disorder with depressed mood).
* Meet the study working definition of burnout which will involve a score on the emotional exhaustion subscale (≥ 27) and a 'high' score on one other subscale (either depersonalization ≥ 13 or personal accomplishment ≤ 21).
* Not taking regularly scheduled medications to treat depression and/or anxiety, including benzodiazepines, for at least 4 weeks prior to initiation of the study.
* Fluent in English.
* Reading literacy and comprehension sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* ECOG Performance Status < or = 2.
* Have a support person that would be able to escort the subject home on the evening of the psilocybin dosing session. The use of ride services will not be permitted (e.g., Uber, Lift, taxi, etc.)
* Adequate liver function as defined as:
* Total Bilirubin < 1.5x institutional upper limit of normal (ULN) unless elevated bilirubin is related to Gilbert's Syndrome.
* AST(SGOT)/ALT(SGPT) <3 x institutional ULN
* For female subjects: Negative pregnancy test and agreement to use highly effective contraception or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause.
* For male subjects: agree to condom use during intercourse for 24 hours post-psilocybin dose.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, ondansetron, cannabis, and non-routine PRN medications within 24 hours of the psilocybin administration. Exceptions include daily use of caffeine, nicotine, and opioid pain medication.
* Agree that for one week preceding the psilocybin session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Agree not to use nicotine for at least 2 hours before the psilocybin administration and for the duration of the psilocybin session.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of the psilocybin session. If the subject does not routinely consume caffeinated beverages, he or she must agree not to do so on the day of psilocybin administration.
* Subjects requiring opioid use for pain are on a stable pain management regimen. Long-acting opioid medications (e.g., oxycodone sustained-release, morphine sustained release) will be allowed if the last dose occurred at least 6 hours before psilocybin administration; such medication will not be taken again until at least 6 hours after psilocybin administration.

Exclusion Criteria:

Yes/No Eligibility Questions (Response of "yes" = subject ineligible)

* Prior systemic antidepressants, antipsychotic, or anxiolytic medication within four weeks prior to study initiation.
* Personal history or first- or second-degree relatives with schizophrenia, bipolar affective disorder, delusional disorder, schizoaffective disorder, psychosis, or other psychotic spectrum illness as determined by patient report and chart review.
* Current or history within the last two years of meeting DSM-V criteria of substance use disorder (excluding caffeine and nicotine). Current substance use disorders may be identified through the drug urine screening test as determined by patient report and chart review.
* Currently meeting DSM-V criteria for Dissociative Disorder, or other psychiatric conditions judged to be incompatible with the establishment of rapport or safe exposure to psilocybin as determined by patient report and chart review.
* Currently meeting DSM-V criteria for Cluster B Personality Disorder as determined by patient report and chart review.
* Severe depression requiring immediate standard-of-care treatment (e.g., hospitalization).
* Suicidal ideation over the past month as assessed as a yes to question 3, 4, or 5 on the Columbia-Suicide Severity Rating Scale, Suicidal Ideation section
* Cancer with known CNS involvement, previously treated brain metastasis, or other major CNS disease.
* Employment as house staff/residents
* The subject has uncontrolled significant intercurrent or recent illness including, but not limited to, the following conditions:
* Cardiovascular disorders: Congestive heart failure, including all New York Heart Association Classes.
* Angina pectoris, cardiac hypertrophy, cardiac ischemia, myocardial infarction
* Uncontrolled hypertension at the time of enrollment (BP>140 systolic or 90 diastolic), coronary artery disease, artificial heart valve
* Prolonged or congenital long QT syndrome (>450 ms), serious cardiac arrhythmias, tachycardia, a clinically significant screening ECG abnormality
* Renal insufficiency as defined as creatinine clearance < 40 mL/min calculated by Cockcroft-Gault formula
* Hepatic disorders: Active infection including hepatitis B (known positive HBV surface antigen (HBsAg) result) or hepatitis C.
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [patients may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Known prior severe hypersensitivity to investigational product or any component in its formulations (NCI CTCAE v5.0 Grade > 3).
* Subjects taking prohibited medications. A washout period of prohibited medications for a period of at least five half-lives should occur prior to study registration.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of MBSR + PAP vs. MBSR alone in reducing symptoms of depression, as measured by the QIDS-SR-16 | 6 months
  Efficacy will be assessed through mean reduction in QIDS-SR-16 scores at 2-weeks post intervention with between-group comparison. To understand longitudinal effects, the investigators will gather data to 6 months post intervention for both arms. Participants will be screened for eligibility with the PHQ-9 with a cut-off score of ≥ 8 required for enrollment.

SECONDARY OUTCOMES:
Effect of MBSR + PAP vs. MBSR alone on participant reported symptoms of burnout as measured by the Maslach Burnout Inventory, MBI-HSS(MP). | Study enrollment to 2 weeks post completion of intervention as well as 6 months post intervention.
  Mean change in MBI-HSS(MP) scores from baseline to 2 weeks and 6 months post intervention with between-group comparison.
Effect of MBSR+PAP vs. MBSR alone on symptoms of demoralization | Study enrollment to 2 weeks post completion of intervention
  Change in scores on the Demoralization II Scale from baseline to 2-weeks post completion of intervention.
Effect of MBSR + PAP vs. MBSR alone on symptoms of post-traumatic stress | Study enrollment to 2 weeks post completion of intervention
  Change in PCL-5 PTSD Checklist scores from baseline to 2 weeks post intervention
Effect of MBSR + PAP vs. MBSR alone on participant reported quality of life. | Study enrollment to 2 weeks post intervention
  The change in the McGill Quality of Life Questionnaire (MQOL) score from baseline to two weeks post-completion of intervention.
Effect of MBSR + PAP vs. MBSR alone on measures of connectedness to self, other, and world | Study enrollment to 2 weeks post intervention
  The change in score on the Watts' Connectedness Scale (WCS) scale from baseline to two weeks post-¬completion of the intervention.
Storyline Health Integrative Assessment | Study enrollment to 2 weeks and 6 months post intervention
  Investigators will deploy the Storyline Integrative Assessment to narrow in on specific feature selection in small cohorts of patients with deep AI phenotyping to identify behavioral phenotype predictors of burnout, which is heterogeneously characterized. This will be administered to both study arms at baseline, at the primary outcome point (2 weeks post intervention on both study arms), and at 6 months post intervention.
  Investigators will deploy Storyline technology to narrow in on specific feature selection using deep AI phenotyping to identify phenotypical predictors of treatment response to both MBSR as well as MBSR+PAP to better characterize factors that predict response to both interventions, which may inform future research. This will be administered to both study arms at baseline, at the primary outcome point (2 weeks post intervention on both study arms), and at 6 months post intervention.
State and Trait Mindfulness | Study enrollment to 2 weeks post intervention.
  Assess the effect of MBSR + PAP vs. MBSR on measures of state and trait mindfulness using the Five Facet Mindfulness Questionnaire (FFMQ) and the Toronto Mindfulness Scale (TMS).

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Mental Health Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis BR, Hendrick J, Byrne K, Odette M, Wu C, Garland EL. Psilocybin-assisted group psychotherapy and mindfulness-based stress reduction for frontline healthcare provider COVID-19-related depression and burnout: A randomized controlled trial. PLoS Med. 2025 Sep 19;22(9):e1004519. doi: 10.1371/journal.pmed.1004519. eCollection 2025 Sep. PMID 40972137
- [Derived] Lewis BR, Garland EL, Byrne K, Durns T, Hendrick J, Beck A, Thielking P. HOPE: A Pilot Study of Psilocybin Enhanced Group Psychotherapy in Patients With Cancer. J Pain Symptom Manage. 2023 Sep;66(3):258-269. doi: 10.1016/j.jpainsymman.2023.06.006. Epub 2023 Jun 10. PMID 37302533